CLINICAL TRIAL: NCT06868953
Title: Use of the Combination of Sumatriptan and Naproxen in the Acute Treatment of Migraine: Real World Evidence Study
Acronym: SMART
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: IRCCSSanRaffaeleRoma
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Migraine
Keywords: migraine attack
MeSH Terms: conditions — Migraine Disorders | interventions — Naproxen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Migraineurs with >4 monthly migraine days: Consecutive adults with episodic migraine (EM) or chronic migraine (CM) with more than 4 days of migraine per month who attend Headache Centers and have been prescribed at least one dose of sumatriptan 85 mg in combination with naproxen 500 mg for the acute treatment of migraine will be enrolled.
  Interventions: Drug: combination of sumatriptan 85 mg and naproxen 500 mg

INTERVENTIONS:
Drug: combination of sumatriptan 85 mg and naproxen 500 mg — combination of sumatriptan 85 mg and naproxen 500 mg

SUMMARY:
This is a multicenter, observational, prospective, real-life study that will be conducted at Headache Centers, aimed at confirming the efficacy and safety of the combination of sumatriptan 85 mg with naproxen 500 mg. The combination of sumatriptan 85 mg and naproxen sodium 500 mg is indicated for the acute treatment of migraine attacks, with or without aura, in adult patients for whom sumatriptan monotherapy is insufficient. In two randomized studies, the sumatriptan/naproxen sodium combination demonstrated significantly greater efficacy (65% of participants-n=1461-reported pain freedom at 2 hours) compared to sumatriptan alone (55%), naproxen sodium alone (44%), or placebo (28%) when used as a late therapy for a single migraine episode in adults. Similar results were observed in a second study (n=1495), with 57% of participants achieving pain freedom within 2 hours after taking the sumatriptan/naproxen sodium combination, outperforming both sumatriptan monotherapy (50%) and naproxen sodium monotherapy (43%), as well as placebo (29%). This superiority was further assessed through sustained pain freedom over 24 hours, with an efficacy of 23-25% in participants treated with the sumatriptan/naproxen combination compared to placebo (7-8%; p<0.001 for both studies) and its individual components (sumatriptan monotherapy: 14%-16%; p=0.009 and p<0.001, naproxen sodium monotherapy: 10%).

In four additional randomized studies, the combination was also found to be effective in menstrual migraine and dysmenorrhea, as well as in cases of poor response or intolerance to triptan therapy. In clinical trials, sumatriptan/naproxen sodium was generally well tolerated, with an overall safety profile similar to that of sumatriptan. The most common adverse events were consistent with those expected for sumatriptan and naproxen sodium.

DETAILED DESCRIPTION:
Consecutive episodic or chronic migraine adults (with more than 4 migraine days per month) followed at the Headache Centers and have been prescribed at least one dose of sumatriptan 85 mg in combination with naproxen sodium 500 mg for the acute treatment of migraine will be enrolled.

The collection of demographic and clinical characteristics will be carried out through a direct interview using a detailed, semi-structured questionnaire during the screening/baseline visit, when the prescription of the sumatriptan 85 mg and naproxen sodium 500 mg combination for migraine attacks will be issued. The follow-up visit will occur after 12 weeks (+/-14 days) from the screening/baseline visit, the end of study visit will take place after 24 weeks (+/-14 days) from baseline.

Patients will be provided with paper diaries for the following 12 weeks at screning/baseline visit and at the follow up visit (at week 12). The paper diaries from the previous 12 weeks will be collected will be collected at week 12 and at week 24.

The following questionnaires will be administered:

* Migraine Specific Quality of Life Questionnaire (MSQ)
* Migraine Interictal Burden Scale (MIBS-4)
* Headache Impact Test-6 (HIT-6) were administered at baseline/screening visit, at follow-up visit (at week 12) and at the end of study visit.

Throughout the study, any adverse events will be recorded and managed.

ELIGIBILITY:
Inclusion Criteria:

1. Migraineurs (age ≥18 years, <65 years) with at least 4 migraine days per month according to ICHD-3 criteria who have been prescribed the combination of sumatriptan 85 mg and naproxen 500 mg;
2. Signed informed consent as required;
3. Agreement to comply with all study procedures, including follow-up visits;
4. Use of a contraceptive method by all participants throughout the study duration.

Exclusion Criteria:

1. Age <18 years or >65 years
2. Pregnancy or breastfeeding
3. Poor knowledge of the Italian language
4. Comorbidities with other neurological, cardiovascular, hepatic, respiratory, hematological, or autoimmune diseases, or clinically significant laboratory abnormalities
5. Inability to distinguish migraine attacks from tension-type headaches
6. Migraine characterized by mild attacks or attacks that resolve spontaneously within 2 hours
7. Hemiplegic or basilar migraine
8. Headache with the use of acute medication on more than 10 days per month in each of the 3 months prior to screening
9. Unwillingness to participate in the study -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive adults with episodic migraine (EM) or chronic migraine (CM) with more than 4 days of migraine per month who attend Headache Centers and have been prescribed at least one dose of sumatriptan 85 mg in combination with naproxen 500 mg for the acute treatment of migraine will be enrolled.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
2 hour-pain freedom | 2 hours after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Percentage of patients reporting complete pain relief within 2 hours after taking the combination of sumatriptan 85 mg and naproxen 500 mg (2h-pain freedom).

SECONDARY OUTCOMES:
1 hour-pain freedom | 1 hour after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Percentage of patients reporting complete pain relief within 1 hour after taking the combination of sumatriptan 85 mg and naproxen 500 mg (1h-pain freedom).
2 hour-pain relief | 2 hours after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Percentage of patients reporting a 50% reduction in pain intensity within 2 hours after taking the combination of sumatriptan 85 mg and naproxen 500 mg (2h-pain relief)
Disappearence of Most Bothersome Symptom | 2 hours after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Percentage of patients experiencing the disappearance of the Most Bothersome Symptom (MBS: the accompanying symptom of the attack considered most disabling by the patient) within 2 hours after taking the combination tablet of sumatriptan 85 mg/naproxen 500 mg.
Presence or absence of associated symptoms (nausea, vomiting, photophobia, or phonophobia) | 1-48 hours after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Presence or absence of associated symptoms (nausea, vomiting, photophobia, or phonophobia) at predefined time intervals of 1, 2, 3, 4, 6, 8, 24, and 48 hours.
24 hour-sustained pain freedom | 24 hours after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Percentage of patients experiencing complete pain relief within 2 hours after taking the combination of sumatriptan 85 mg and naproxen 500 mg, with sustained benefit in the following 24 hours (24h-sustained pain freedom).
24 hour sustained pain relief | 24 hours after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Percentage of patients experiencing a 50% reduction in pain intensity within 2 hours after taking the combination of sumatriptan 85 mg and naproxen 500 mg, with sustained benefit in the following 24 hours (24h-sustained pain relief).
headache recurrence | 2 hours after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Definition of the moment of possible migraine pain recurrence (headache recurrence), as well as its intensity within 24 and 48 hours following the administration of the medication (limited to patients who experienced pain freedom within 2 hours).
use of rescue medication | 24 hours after taking combination of sumatriptan 85 mg and naproxen 500 mg
  Use of rescue medications and evaluation of the time interval between the first and second dose.
Variation of Migraine Specific Quality of Life Questionnaire score at week 24 | week 24 after taking the first dose of combination of sumatriptan 85 mg and naproxen 500 mg
  Changes in scores of the Migraine Specific Quality of Life Questionnaire administered at week 24 compared to baseline
Variation of Migraine Specific Quality of Life Questionnaire score at week 24 | week 24 after taking the first dose of combination of sumatriptan 85 mg and naproxen 500 mg
  Changes in scores of the Migraine Specific Quality of Life Questionnaire administered at week 24 compared to week 12
Variation of Migraine Interictal Burden Scale score at week 24 | week 24 after taking the first dose of combination of sumatriptan 85 mg and naproxen 500 mg
  Changes in scores of the Migraine Specific Quality of Life Questionnaire administered at week 24 compared to baseline
Variation of Migraine Interictal Burden Scale score at week 24 | week 24 after taking the first dose of combination of sumatriptan 85 mg and naproxen 500 mg
  Changes in score of the Migraine Interictal Burden Scale administered at week 24 compared to week 12
Variation of Headache Impact Test score at week 24 | week 24 after taking the first dose of combination of sumatriptan 85 mg and naproxen 500 mg
  Changes in score of Headache Impact Test scale administered at week 24 compared to baseline
Variation of Headache Impact Test score score at week 24 | week 24 after taking the first dose of combination of sumatriptan 85 mg and naproxen 500 mg
  Changes in score of Headache Impact Test scale administered at week 24 compared to week 12
Patient Global Impression of Change | week 24 after taking the first dose of combination of sumatriptan 85 mg and naproxen 500 mg
  Collection of subjective feedback from the patient regarding their experience with the medication, assessing patient satisfaction, ease of use of the medication, and perceived effectiveness with Patient Global Impression of Change scale
Adverse events occurrence | 48 hours after taking the first dose of combination of sumatriptan 85 mg and naproxen 500 mg
  Definition of the type and number of adverse events occurring within 48 hours of taking the combination of sumatriptan 85 mg and naproxen 500 mg through a specific questionnaire (event details, duration, severity, and actions taken).

REFERENCES:
- [Background] Brandes JL, Kudrow D, Stark SR, O'Carroll CP, Adelman JU, O'Donnell FJ, Alexander WJ, Spruill SE, Barrett PS, Lener SE. Sumatriptan-naproxen for acute treatment of migraine: a randomized trial. JAMA. 2007 Apr 4;297(13):1443-54. doi: 10.1001/jama.297.13.1443. PMID 17405970
- [Background] Allais G, Castagnoli Gabellari I, Rolando S, Benedetto C. Evaluation of the use of sumatriptan-naproxen sodium for menstrual migraine and dysmenorrhea. Expert Rev Neurother. 2011 Oct;11(10):1383-7. doi: 10.1586/ern.11.123. PMID 21955195
- [Background] Smith TR, Sunshine A, Stark SR, Littlefield DE, Spruill SE, Alexander WJ. Sumatriptan and naproxen sodium for the acute treatment of migraine. Headache. 2005 Sep;45(8):983-91. doi: 10.1111/j.1526-4610.2005.05178.x. PMID 16109111
- [Background] Wilcha RJ, Afridi SK, Barbanti P, Diener HC, Jurgens TP, Lanteri-Minet M, Lucas C, Mawet J, Moisset X, Russo A, Sacco S, Sinclair AJ, Sumelahti ML, Tassorelli C, Goadsby PJ. Sumatriptan-naproxen sodium in migraine: A review. Eur J Neurol. 2024 Sep;31 Suppl 2(Suppl 2):e16434. doi: 10.1111/ene.16434. PMID 39318200
- [Background] Mathew NT, Landy S, Stark S, Tietjen GE, Derosier FJ, White J, Lener SE, Bukenya D. Fixed-dose sumatriptan and naproxen in poor responders to triptans with a short half-life. Headache. 2009 Jul;49(7):971-82. doi: 10.1111/j.1526-4610.2009.01458.x. Epub 2009 May 27. PMID 19486178
- [Background] Silberstein S, McDonald SA, Goldstein J, Aurora S, Lener SE, White J, Runken MC, Saiers J, Derosier F, Lipton RB. Sumatriptan/naproxen sodium for the acute treatment of probable migraine without aura: a randomized study. Cephalalgia. 2014 Apr;34(4):268-79. doi: 10.1177/0333102413508242. Epub 2013 Oct 9. PMID 24108307
- [Background] Lipton RB, Dodick DW, Adelman JU, Kaniecki RG, Lener SE, White JD, Nelsen AC. Consistency of response to sumatriptan/naproxen sodium in a placebo-controlled, crossover study. Cephalalgia. 2009 Aug;29(8):826-36. doi: 10.1111/j.1468-2982.2008.01806.x. Epub 2009 Feb 12. PMID 19220307